CLINICAL TRIAL: NCT04579679
Title: An Open-Label Phase 2 Study of Surufatinib in Patients With Neuroendocrine Tumours in Europe
Brief Title: Open-Label Surufatinib in European Patients With NET
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Hutchmed (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-012-00EU1
Record Dates: First submitted 2020-09-23; First posted 2020-10-08 (Actual); Results first posted 2025-07-25 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Neuroendocrine Tumours; Neuroendocrine Tumour of the Lung; Small Intestinal NET
Keywords: VEGF
MeSH Terms: conditions — Neuroendocrine Tumors | interventions — surufatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Surufatinib (Experimental): Cohorts A, B, and C: oral surufatinib 300 mg once daily in treatment cycles of 28 days starting at Cycle 1 Day1
  Cohort D:
  Surufatinib 300 mg once daily in treatment cycles of 28 days starting at Cycle 1 Day and single doses of drug cocktail on Day-2 and Day 15 Cycle 1
  Interventions: Drug: Surufatinib

INTERVENTIONS:
Drug: Surufatinib — Surufatinib 300 mg oral once daily
  Other Names: HMPL-012, sulfatinib

SUMMARY:
This is a Phase 2, open-label, multi-centre study of surufatinib in patients with low to intermediate grade (Grade 1 or Grade 2), well-differentiated neuroendocrine tumours (NETs).

DETAILED DESCRIPTION:
This is a Phase 2, open-label, multi-centre study of surufatinib in patients with low- to intermediate-grade (Grade 1 or Grade 2), well-differentiated NETs.

The study will enroll 4 cohorts of varying NETs, as follows:

* Cohort A - NET of lung origin
* Cohort B - NET of small bowel origin
* Cohort C - NET of non-small bowel, non-pancreas, and non-lung origin
* Cohort D - NET of any origin (DDI substudy)

All patients will be treated with oral surufatinib 300 mg QD in treatment cycles of 28 days starting on Cycle 1 Day 1.

ELIGIBILITY:
Key Inclusion Criteria:

1. Has histologically or cytologically documented, locally advanced, or metastatic NET and has progressed on at least 1 prior line of therapy, but no more than 3 therapies;
2. Has radiologic evidence of progressive tumour within 12 months of study enrolment
3. Is willing and able to provide informed consent
4. Is ≥18 years of age
5. Has measurable lesions according to RECIST Version 1.1
6. Has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
7. Female patients of childbearing potential and male patients with partners of childbearing potential agree to use a highly effective form(s) of contraception

Key Exclusion Criteria:

1. Has an AE due to previous anti-tumour therapy that has not recovered to ≤CTCAE Grade 1, except alopecia and peripheral neurotoxicity with ≤CTCAE Grade 2 caused by platinum chemotherapy
2. Major surgery within previous 4 weeks or radiation therapy within 2 weeks prior to the start of treatment.
3. Prior VEGF/VEGFR-targeted therapy
4. Uncontrollable hypertension, defined as systolic blood pressure ≥140 mmHg and/or diastolic blood pressure ≥90 mmHg, despite antihypertensive medication
5. Gastrointestinal disease or condition within 6 months prior to first dose
6. Has a history or presence of a serious haemorrhage (>30 mL within 3 months) or haemoptysis (>5 mL blood within 4 weeks) within 6 months of first dose of study drug.
7. Clinically significant cardiovascular disease.
8. Brain metastases and/or spinal cord compression untreated with surgery and/or radiotherapy, and without clinical imaging evidence of stable disease (SD) for 14 days or longer; patients requiring steroids within 4 weeks prior to start of study treatment will be excluded.
9. A high risk of bleeding at screening due to tumour invasion into major vessels, such as pulmonary artery, the superior vena cava, or the inferior vena cava, as determined by investigators.
10. Has arterial thrombosis or deep venous thrombosis within 6 months prior to first dosing, or thromboembolic events (including stroke and/or transient ischaemic attack) within 12 months.
11. Has a clinically meaningful ongoing infection (eg, requiring intravenous treatment with anti-infective therapy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2021-08-13 (Actual); Primary Completion 2024-09-06 (Actual); Study Completion 2024-10-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Schelman, MD, PhD, Study Director — Hutchmed
Locations (23):
- United States (5):
  - University of Alabama, Birmingham (UAB), Birmingham, Alabama
  - University of California Irvine Medical Center UCIMC - H.H. Chao Comprehensive Digestive Disease Center CDDC, Orange, California
  - Emory University, Winship Cancer Institute, Atlanta, Georgia
  - Stony Brook Cancer Center, Stony Brook, New York
  - Houston Methodist, Houston, Texas
- France (2):
  - CHU Bordeaux, Pessac
  - Institut Gustave Roussy, Villejuif
- Germany (3):
  - Charite Universitatsmedizin Berlin, Berlin
  - Universitaetsklinikum Erlangen, Erlangen
  - Universitatsklinikum Essen, Klinik fur Endokrinologie, Essen
- Italy (4):
  - Azienda Universitaria Ospedaliera Consorziale - Policlinico Bari, Bari
  - ASST-Spedali Civili di Brescia, Brescia
  - Universita degli Studi di Firenze - Azienda Ospedaliero Universitaria Careggi (AOUC), Florence
  - Istituto Europeo di Oncologia, Milan
- Norway (2):
  - Haukeland University Hospital, Bergen
  - Oslo University Hospital Rikshospitalet, Oslo
- Spain (5):
  - Institut Catala d'Oncologis (ICO) - Hospital Duran i Reynals, Barcelona
  - Hospital Vall Hebron, Barcelona
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Virgen del Rocio, Seville
- United Kingdom (2):
  - Sarah Cannon Research Institute, London
  - Christie Hospital, Manchester

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This Phase 2, multicenter, open-label study was conducted in patients with locally advanced or metastatic low to intermediate grade (Grade 1 or Grade 2), well-differentiated neuroendocrine tumors (NETs).
Pre-assignment Details: The study enrolled patients in 4 cohorts of varying NETs as follows:
  * Cohort A - NET of lung origin (NET, lung)
  * Cohort B - NET of small bowel origin (NET, small bowel)
  * Cohort C - NET of non-small bowel, non-pancreas, and non-lung origin (NET, other)
  * Cohort D - NET of any origin/drug-drug interaction sub-study (NET, any)
  The study was terminated early based on the strategic re-evaluation of the clinical development program for surufatinib and not due to any safety concerns.
Groups:
- Cohort A (NET, Lung): Patients with NET of lung origin received surufatinib 300 milligrams (mg) orally once daily (QD) in treatment cycles of 28 days starting on Cycle (C)1 Day (D)1 until disease progression, death, unacceptable toxicity, withdrawal of consent or lost to follow-up.
- Cohort B (NET, Small Bowel): Patients with NET of small bowel origin received surufatinib 300 mg orally QD in treatment cycles of 28 days starting on C1D1 until disease progression, death, unacceptable toxicity, withdrawal of consent or lost to follow-up.
- Cohort C (NET, Other): Patients with NET of non-small bowel, non-pancreas, and non-lung origin received surufatinib 300 mg orally QD in treatment cycles of 28 days starting on C1D1 until disease progression, death, unacceptable toxicity, withdrawal of consent or lost to follow-up.
- Cohort D (NET, Any): Patients with NET of any origin received a single dose of drug cocktail (midazolam 2.5 mg, fexofenadine 30 mg and rosuvastatin 10 mg) on Day -2 followed by surufatinib 300 mg orally QD from C1D1 to C1D14. On C1D15, a single dose of surufatinib 300 mg and a single dose of drug cocktail as above was administered. Patients received surufatinib 300 mg orally QD from C1D16 until disease progression, death, unacceptable toxicity, withdrawal of consent or lost to follow-up.
Period: Overall Study
Arm/Group | Cohort A (NET, Lung) | Cohort B (NET, Small Bowel) | Cohort C (NET, Other) | Cohort D (NET, Any)
Started | 20 | 32 | 20 | 6
Completed | 0 | 1 | 0 | 2
Not Completed | 20 | 31 | 20 | 4
Not completed — New Antitumor Therapy | 6 | 4 | 7 | 0
Not completed — Withdrawal of Consent | 1 | 1 | 2 | 4
Not completed — Death | 2 | 2 | 2 | 0
Not completed — Adverse Event | 0 | 4 | 0 | 0
Not completed — Disease Progression | 9 | 13 | 7 | 0
Not completed — Physician Decision | 0 | 0 | 1 | 0
Not completed — Study Terminated by Sponsor | 2 | 7 | 1 | 0

BASELINE CHARACTERISTICS:
Population: The safety analysis set included all patients who received at least 1 dose of surufatinib.
Groups:
- Cohort A (NET, Lung): Patients with NET of lung origin received surufatinib 300 mg orally QD in treatment cycles of 28 days starting on C1D1 until disease progression, death, unacceptable toxicity, withdrawal of consent or lost to follow-up.
- Total: Total of all reporting groups
Arm/Group | Cohort A (NET, Lung) | Cohort B (NET, Small Bowel) | Cohort C (NET, Other) | Cohort D (NET, Any) | Total
Number analyzed (Participants) | 20 | 32 | 20 | 6 | 78
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.5 (12.77) | 62.1 (10.44) | 57.3 (15.52) | 63.5 (7.40) | 61.3 (12.37)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 20 | 9 | 4 | 40
  Male | 13 | 12 | 11 | 2 | 38
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 3 | 0 | 0 | 3
  Not Hispanic or Latino | 15 | 26 | 13 | 6 | 60
  Unknown or Not Reported | 5 | 3 | 7 | 0 | 15
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 0 | 1
  Black or African American | 0 | 0 | 0 | 3 | 3
  White | 15 | 28 | 13 | 3 | 59
  Not Reported | 4 | 1 | 7 | 0 | 12
  Other | 0 | 1 | 0 | 0 | 1
  Missing | 1 | 1 | 0 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Disease Control Rate (DCR)
Description: The DCR was defined as the percentage of patients who achieved a best overall response (BOR) of complete response (CR), partial response (PR) or stable disease (SD) as determined by the Investigator using Response Evaluation Criteria in Solid Tumors (RECIST) version (v)1.1. The CR was defined as disappearance of all target lesions. The PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum of diameters. SD was defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (PD), taking as reference the smallest sum on study.
Time Frame: RECIST assessments performed at screening (within 28 days before start of study drug), every 8 weeks for the first 24 weeks from C1D1, then every 12 weeks thereafter until the occurrence of disease progression, up to approximately 36 months
Population: The efficacy analysis set included all patients who received at least 1 dose of surufatinib and had at least 1 post-baseline tumor assessment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort A (NET, Lung) | Cohort B (NET, Small Bowel) | Cohort C (NET, Other) | Cohort D (NET, Any)
Number analyzed (Participants) | 20 | 31 | 19 | 5
percentage of participants | 95.0 [75.1 to 99.9] | 90.3 [74.2 to 98.0] | 89.5 [66.9 to 98.7] | 100 [47.8 to 100]

2. Secondary Outcome: Plasma Concentrations of Surufatinib
Description: Blood samples were collected at specified timepoints to obtain plasma concentrations of surufatinib at steady state on Cycle 1 Day 15.
Time Frame: Cohorts A, B and C: Pre-dose and 1, 2, 3, 4 hours post-dose on Cycle 1 Day 15; Cohort D: Pre-dose and 30 minutes, 1, 2, 3, 4, 5, 6, 8 and 10 hours post-dose on Cycle 1 Day 15
Population: The pharmacokinetic (PK) analysis set included all patients who received at least 1 dose of the study drug and had at least 1 measurable plasma concentration data point for at least 1 PK analyte without protocol violations or events with potential to affect the PK concentration. Only those participants with data collected at specified timepoints are reported.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram/milliliter
Arm/Group | Cohort A (NET, Lung) | Cohort B (NET, Small Bowel) | Cohort C (NET, Other) | Cohort D (NET, Any)
Number analyzed (Participants) | 17 | 29 | 18 | 6
nanogram/milliliter
  Pre-dose: number analyzed (Participants) | 17 | 25 | 18 | 6
  Pre-dose | 73.123 (70.1) | 57.593 (136.8) | 49.258 (54.7) | 28.913 (130.5)
  30 minutes post-dose: number analyzed (Participants) | 0 | 0 | 0 | 6
  30 minutes post-dose |  |  |  | 50.439 (190.5)
  1 hour post-dose: number analyzed (Participants) | 17 | 29 | 15 | 6
  1 hour post-dose | 130.456 (118.3) | 96.163 (115.2) | 101.464 (125.6) | 129.719 (303.6)
  2 hours post-dose: number analyzed (Participants) | 17 | 27 | 18 | 6
  2 hours post-dose | 234.498 (122.1) | 174.799 (138.1) | 194.654 (80.5) | 321.942 (99.9)
  3 hours post-dose | 287.237 (95.0) | 250.348 (101.8) | 245.379 (55.1) | 477.653 (118.6)
  4 hours post-dose: number analyzed (Participants) | 17 | 28 | 17 | 6
  4 hours post-dose | 293.236 (85.6) | 268.619 (65.9) | 232.657 (42.6) | 389.597 (102.8)
  5 hours post-dose: number analyzed (Participants) | 0 | 0 | 0 | 6
  5 hours post-dose |  |  |  | 357.045 (105.4)
  6 hours post-dose: number analyzed (Participants) | 0 | 0 | 0 | 6
  6 hours post-dose |  |  |  | 280.691 (105.2)
  8 hours post-dose: number analyzed (Participants) | 0 | 0 | 0 | 6
  8 hours post-dose |  |  |  | 202.345 (102.7)
  10 hours post-dose: number analyzed (Participants) | 0 | 0 | 0 | 4
  10 hours post-dose |  |  |  | 174.079 (84.1)

3. Secondary Outcome: Number of Patients With Potentially Clinically Significant Corrected QT Interval (QTc) During Treatment
Description: The QT interval data was corrected for heart rate using 2 correction methods (Fridericia - QTcF and Bazett - QTcB). The treatment period was defined as the period from first administration of study drug up 30 days after last administration. msec=milliseconds, IFB=increase from baseline.
Time Frame: From the first dose of study drug (Day 1) up to 30 days after last dose of study drug, approximately 33 months
Population: The safety analysis set included all patients who received at least 1 dose of surufatinib. Only those patients with data collected are reported.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A (NET, Lung) | Cohort B (NET, Small Bowel) | Cohort C (NET, Other) | Cohort D (NET, Any)
Number analyzed (Participants) | 19 | 31 | 19 | 6
Participants
  QTcF: >450 msec to <=480 msec: number analyzed (Participants) | 19 | 31 | 18 | 6
  QTcF: >450 msec to <=480 msec | 0 | 2 | 0 | 2
  QTcF: >480 msec to <=500 msec: number analyzed (Participants) | 19 | 31 | 18 | 6
  QTcF: >480 msec to <=500 msec | 0 | 4 | 1 | 0
  QTcF: >500 msec: number analyzed (Participants) | 19 | 31 | 18 | 6
  QTcF: >500 msec | 0 | 0 | 0 | 1
  QTcF: IFB >30 msec to <=60 msec: number analyzed (Participants) | 19 | 31 | 18 | 6
  QTcF: IFB >30 msec to <=60 msec | 4 | 2 | 1 | 1
  QTcF: IFB >60 msec: number analyzed (Participants) | 19 | 31 | 18 | 6
  QTcF: IFB >60 msec | 0 | 2 | 0 | 1
  QTcB: >450 msec to <=480 msec | 3 | 6 | 3 | 4
  QTcB: >480 msec to <=500 msec | 0 | 1 | 0 | 1
  QTcB: >500 msec | 0 | 1 | 1 | 1
  QTcB: IFB >30 msec to <=60 msec | 2 | 7 | 4 | 1
  QTcB: IFB >60 msec | 1 | 2 | 0 | 1

4. Secondary Outcome: Objective Response Rate (ORR)
Description: The ORR was defined as the percentage of patients with a BOR of CR or PR as determined by the Investigator using RECIST v1.1. The CR was defined as disappearance of all target lesions. The PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum of diameters.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort A (NET, Lung) | Cohort B (NET, Small Bowel) | Cohort C (NET, Other) | Cohort D (NET, Any)
Number analyzed (Participants) | 20 | 31 | 19 | 5
percentage of participants | 15.0 [3.2 to 37.9] | 16.1 [5.5 to 33.7] | 5.3 [0.1 to 26.0] | 20.0 [0.5 to 71.6]

5. Secondary Outcome: Time to Response (TTR)
Description: The TTR was defined as the time from the start of study drug until the date of first documented objective response, either CR or PR (whichever was recorded first) according to RECIST v.1.1 for responders only. The CR was defined as disappearance of all target lesions. The PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum of diameters.
Time Frame: as for outcome 1
Population: The efficacy analysis set included all patients who received at least 1 dose of surufatinib and had at least 1 post-baseline tumor assessment. Only those patients who achieved CR or PR (responders) were included in the analysis.
Measure: Median (Full Range); unit: months
Arm/Group | Cohort A (NET, Lung) | Cohort B (NET, Small Bowel) | Cohort C (NET, Other) | Cohort D (NET, Any)
Number analyzed (Participants) | 3 | 5 | 1 | 1
months | 2.1 [1.6 to 5.3] | 3.7 [1.8 to 14.2] | 11.1 [11.1 to 11.1] | 13.6 [13.6 to 13.6]

6. Secondary Outcome: Duration of Response (DOR)
Description: The DoR was defined as the time from the first time that the objective response reached CR or PR, whichever came first (and later confirmed), until the occurrence of PD or death. The CR was defined as disappearance of all target lesions. The PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum of diameters. The PD was defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (nadir), including baseline. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 millimeters. The appearance of 1 or more new lesions was also considered progression.
Time Frame: as for outcome 1
Population: as for outcome 5
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort A (NET, Lung) | Cohort B (NET, Small Bowel) | Cohort C (NET, Other) | Cohort D (NET, Any)
Number analyzed (Participants) | 3 | 5 | 1 | 1
months | 16.9 [8.6 to NA] — NA indicates that upper limit of confidence interval (CI) was not estimable due to insufficient number of patients with events at study closure. | 15.4 [3.7 to NA] — NA indicates that upper limit of CI was not estimable due to insufficient number of patients with events at study closure. | 5.6 [NA to NA] — NA indicates that upper and lower limits of CI could not be calculated for 1 patient. | NA [NA to NA] — NA indicates that median, upper and lower limit of CI was not estimable due to insufficient number of patients with events at study closure.

7. Secondary Outcome: Progression-Free Survival (PFS)
Description: The PFS was defined as the time from the start of study drug until the first objective PD as defined by RECIST v1.1 or death, whichever came first. The PD was defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (nadir), including baseline. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 millimeters. The appearance of 1 or more new lesions was also considered progression.
Time Frame: as for outcome 1
Population: The safety analysis set included all patients who received at least 1 dose of surufatinib.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort A (NET, Lung) | Cohort B (NET, Small Bowel) | Cohort C (NET, Other) | Cohort D (NET, Any)
Number analyzed (Participants) | 20 | 32 | 20 | 6
months | 10.2 [5.4 to 16.6] | 19.2 [8.3 to NA] — NA indicates that upper limit of CI was not estimable due to insufficient number of patients with events at study closure. | 11.4 [5.7 to 16.7] | 9.8 [7.2 to NA] — NA indicates that upper limit of CI was not estimable due to insufficient number of patients with events at study closure.

8. Secondary Outcome: Cohort D: Geometric Least Squares (LS) Mean Ratio of Cytochrome P450 (CYP3A4), P-glycoprotein (P-gp) and Breast Cancer Resistance Protein (BCRP) Substrates at Cycle 1 Day 15 to Baseline
Description: Participants were administered midazolam, fexofenadine and rosuvastatin (as part of the drug cocktail) as a single dose on Day -2 (without surufatinib) and on Cycle 1 Day 15 (with surufatinib). Separate blood samples were collected for measurement of plasma concentrations of each probe substrate and surufatinib. Probe substrate of midazolam was CYP3A4, fexofenadine was P-gp and rosuvastatin was BCRP. Ratio of LS Mean for maximum plasma concentration (Cmax), area under the plasma concentration-time curve from time 0 to time of last measurable concentration (AUC0-t) and area under the plasma concentration-time curve from time 0 to infinity (AUC0-inf) are presented as Cycle 1 Day 15/Day -2.
Time Frame: Baseline (Day -2) and Cycle 1 Day 15
Population: The PK evaluable population included all patients who received at least 1 dose of the study drug and had sufficient concentration data to derive at least 1 PK parameter.
Measure: Number (90% Confidence Interval); unit: Ratio of geometric LS mean
Arm/Group | Cohort D (NET, Any)
Number analyzed (Participants) | 6
Ratio of geometric LS mean
  Midazolam (CYP3A4 substrate), Cmax | 1.69 [1.20 to 2.39]
  Midazolam (CYP3A4 substrate), AUC0-t | 1.70 [1.14 to 2.52]
  Midazolam (CYP3A4 substrate), AUC0-inf | 1.71 [1.16 to 2.53]
  Fexofenadine (P-gp substrate), Cmax | 2.03 [1.51 to 2.75]
  Fexofenadine (P-gp substrate), AUC0-t | 2.12 [1.65 to 2.73]
  Fexofenadine (P-gp substrate), AUC0-inf | 2.14 [1.64 to 2.78]
  Rosuvastatin (BCRP substrate), Cmax | 2.23 [1.59 to 3.14]
  Rosuvastatin (BCRP substrate), AUC0-t | 2.13 [1.31 to 3.48]
  Rosuvastatin (BCRP substrate), AUC0-inf | 2.23 [1.23 to 4.01]

9. Secondary Outcome: Number of Patients With Treatment-emergent Adverse Events (TEAEs) and Treatment-emergent Serious Adverse Events (TESAEs)
Description: An AE is any untoward medical occurrence in a clinical study patient temporally associated with the use of a study drug, whether or not considered related to the drug. An SAE was an AE that resulted in any of the following outcomes: death; was life threatening; required inpatient hospitalization or prolongation of existing hospitalization; resulted persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions; a congenital anomaly/birth defect or was any important medical event. TEAEs were defined as any AEs that started or worsened in severity on or after the first administration date of study drug and no later than 30 (+7) days after the last administration date of study drug or initiation of new anti-tumor therapy (whichever occurred first).
Time Frame: From the first dose of study drug (Day 1) up to 30 days after last dose of study drug, approximately 33 months
Population: The safety analysis set included all patients who received at least 1 dose of surufatinib.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A (NET, Lung) | Cohort B (NET, Small Bowel) | Cohort C (NET, Other) | Cohort D (NET, Any)
Number analyzed (Participants) | 20 | 32 | 20 | 6
Participants
  TEAEs | 20 | 32 | 20 | 6
  TESAEs | 4 | 12 | 8 | 2

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the first dose of study drug (Day 1) up to 30 days after last dose of study drug, approximately 33 months. Deaths were collected from screening (Day -28) up to end of follow-up, approximately 36 months
Description: The safety analysis set included all patients who received at least 1 dose of surufatinib.
Arm/Group | Cohort A (NET, Lung) | Cohort B (NET, Small Bowel) | Cohort C (NET, Other) | Cohort D (NET, Any)
All-Cause Mortality (participants affected / at risk) | 2/20 | 2/32 | 2/20 | 0/6
Serious Adverse Events (participants affected / at risk) | 4/20 | 12/32 | 8/20 | 2/6
Other Adverse Events (participants affected / at risk) | 20/20 | 32/32 | 20/20 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A (NET, Lung) (N=20) | Cohort B (NET, Small Bowel) (N=32) | Cohort C (NET, Other) (N=20) | Cohort D (NET, Any) (N=6)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Large intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Atrioventricular block (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
General physical health deterioration (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Biliary obstruction (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiac function test abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal artery dissection (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Renal infarct (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Asthmatic crisis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertensive emergency (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Multisystem inflammatory syndrome (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Balance disorder (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A (NET, Lung) (N=20) | Cohort B (NET, Small Bowel) (N=32) | Cohort C (NET, Other) (N=20) | Cohort D (NET, Any) (N=6)
Asthenia (General disorders) | 14 (49) | 20 (47) | 13 (22) | 0 (0)
Pyrexia (General disorders) | 6 (11) | 7 (12) | 4 (4) | 0 (0)
Fatigue (General disorders) | 1 (1) | 10 (17) | 1 (6) | 3 (4)
Oedema peripheral (General disorders) | 3 (4) | 7 (9) | 3 (3) | 0 (0)
Mucosal inflammation (General disorders) | 2 (3) | 2 (3) | 1 (1) | 0 (0)
Influenza like illness (General disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Oedema (General disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 11 (20) | 22 (82) | 13 (24) | 2 (4)
Nausea (Gastrointestinal disorders) | 5 (7) | 10 (30) | 4 (6) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 2 (4) | 11 (23) | 3 (3) | 0 (0)
Vomiting (Gastrointestinal disorders) | 6 (8) | 5 (19) | 4 (6) | 1 (2)
Constipation (Gastrointestinal disorders) | 2 (3) | 4 (4) | 5 (6) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 3 (3) | 3 (3) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 2 (3) | 3 (3) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 2 (4) | 1 (1) | 2 (2) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 2 (5) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 14 (32) | 16 (41) | 15 (35) | 3 (4)
Flushing (Vascular disorders) | 1 (3) | 2 (2) | 2 (2) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 2 (3) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 3 (6) | 8 (14) | 2 (3) | 0 (0)
Blood bilirubin increased (Investigations) | 5 (12) | 2 (5) | 4 (11) | 1 (1)
Alanine aminotransferase increased (Investigations) | 2 (2) | 6 (13) | 2 (3) | 0 (0)
Weight decreased (Investigations) | 5 (5) | 2 (2) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 3 (5) | 2 (4) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 3 (3) | 1 (2) | 2 (4) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 3 (3) | 0 (0) | 1 (2)
Amylase increased (Investigations) | 3 (3) | 0 (0) | 0 (0) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 1 (2) | 2 (4) | 1 (2) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Blood thyroid stimulating hormone increased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Bilirubin conjugated increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood pressure increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Troponin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (6) | 9 (17) | 4 (8) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (6) | 4 (7) | 4 (6) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 3 (3) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (3) | 1 (2) | 2 (4) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 4 (6) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (3) | 2 (2)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (4) | 2 (2) | 0 (0) | 0 (0)
Torticollis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 5 (7) | 6 (20) | 7 (14) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 3 (3) | 2 (2) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 2 (2) | 3 (3)
Hyperuricaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (3) | 1 (1) | 1 (1)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 3 (9) | 0 (0) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 3 (3) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (4)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 1 (2) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 3 (3) | 11 (16) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 5 (5) | 3 (4) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (2) | 3 (3) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 1 (2) | 2 (2) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 7 (20) | 7 (15) | 6 (10) | 2 (4)
Haematuria (Renal and urinary disorders) | 3 (3) | 2 (4) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (9) | 1 (2) | 4 (4) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (4) | 1 (1) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (4) | 2 (2) | 2 (2) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 1 (2) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (5) | 2 (2) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 4 (4) | 0 (0) | 1 (1)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (5) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Rash macular (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 6 (8) | 4 (5) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 3 (3) | 1 (1) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 1 (1) | 4 (7) | 0 (0)
Dysgeusia (Nervous system disorders) | 1 (1) | 2 (4) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 2 (3) | 1 (2) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 5 (8) | 3 (8) | 1 (2)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Hypothyroidism (Endocrine disorders) | 2 (4) | 8 (8) | 0 (0) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
Thyroid pain (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 5 (5) | 0 (0) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 (1) | 2 (3) | 0 (0) | 1 (3)
Hypertransaminasaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diplopia (Eye disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Acute vestibular syndrome (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Erectile dysfunction (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Genital hypoaesthesia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Heavy menstrual bleeding (Reproductive system and breast disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscle rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tooth fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sunburn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Based upon the strategic reevaluation of the clinical development program for surufatinib in Europe and the United States (US), the study was terminated. The termination was not based on any concern for patient safety or efficacy relative to surufatinib treatment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2023-12-01): https://cdn.clinicaltrials.gov/large-docs/79/NCT04579679/Prot_000.pdf
  • Statistical Analysis Plan (2024-10-10): https://cdn.clinicaltrials.gov/large-docs/79/NCT04579679/SAP_001.pdf